CLINICAL TRIAL: NCT02522689
Title: Comparison of Success Rates, Complication Rates and Injury to Kidneys of Ultra-mini PCNL and Micro PCNL in the Treatment of Kidney Stones
Brief Title: Comparison of Ultra-mini PCNL and Micro PCNL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Selcuk University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Ozcan Kilic, M.D., Assoc. Prof. Dr., Selcuk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SU-PCNL-UMMP-02
Record Dates: First submitted 2015-08-09; First posted 2015-08-13 (Estimated); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Kidney Stones
Keywords: kidney stone; percutaneous nephrolithotripsy; ultra-mini PCNL; micro PCNL
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultra-mini PCNL (Active Comparator): Endoscopic kidney stone surgery: Patients will undergo ultra-mini percutaneous nephrolithotripsy.
  Interventions: Procedure: Endoscopic kidney stone surgery
- Micro PCNL (Active Comparator): Endoscopic kidney stone surgery: Patients will undergo micro percutaneous nephrolithotripsy.
  Interventions: Procedure: Endoscopic kidney stone surgery

INTERVENTIONS:
Procedure: Endoscopic kidney stone surgery — Ultra-mini PCNL will be performed.
  Arms: Ultra-mini PCNL
Procedure: Endoscopic kidney stone surgery — Micro PCNL will be performed.
  Arms: Micro PCNL

SUMMARY:
It is aimed to evaluate the treatment results, rates of success and complications, and injury given to the kidney by measuring preoperative and postoperative blood and Cystatin C levels in patients with kidney stones smaller than 2 cm who will undergo either ultra-mini percutaneous nephrolithotripsy (PCNL) or micro PCNL.

DETAILED DESCRIPTION:
In this study, the demographic and preoperative data, imaging data, operative data and postoperative follow-up data will be prospectively recorded according to the patient information forms for the patients with kidney stone smaller than 2 cm who will undergo either ultra-mini PCNL or micro PCNL.

A total of 60 (sixty) patients, aging between 18 and 65 years, with similar stone size and location are being planned to be enrolled into the study; and will be prospectively randomized into two groups with a 1:1 ratio, thus 30 (thirty) patients will receive ultra-mini PCNL while 30 (thirty) patients will undergo micro PCNL.

Preoperatively, blood and urine Cystatin C levels will be measured. After the surgery, blood and urine Cystatin C levels at postoperative 12th hour will be recorded. Besides these, classical kidney function tests, namely blood urea and creatinine levels, will be measured preoperatively and postoperatively.

Parameters listed below will be also recorded and evaluated:

1. Preoperative general evaluation data: Age, height, weight, body-mass index, concomitant comorbidities, prescriptions used, history of operation(s), American Society of Anesthesiologists (ASA) score
2. Preoperative urological evaluation data: History of extracorporeal shock wave lithotripsy (ESWL)/PCNL/ureterorenoscopy (URS)/retrograde intrarenal surgery (RIRS)/open surgery, whole blood count, kidney function tests, automatic urine test, urine culture, preoperative imaging modality (KUB, US, CT), number-dimensions-localization-composition of stone(s), existence of hydronephrosis
3. Operative data: Access fluoroscopy duration, total access duration, total fluoroscopy duration, operation duration, use of double-J stent, preoperative complications
4. Number of previous ESWL seance, total duration of ESWL, number of shots during ESWL (if any)
5. Follow-up data: Urethral catheterization time, hospitalization time, need of any other treatment for being stone-free, time to full stone-free, duration to removal of double-J stent, existence of residual stone(s), formation of new stone(s), complications in late period

ELIGIBILITY:
Inclusion Criteria:

* Patients who are planned to undergo PCNL due to kidney stone
* Patients with a kidney stone < 2 cm
* Patients between 18 and 65 years old

Exclusion Criteria:

* Patients with unregulated diabetes mellitus and diabetic nephropathy
* Patients with a blood pressure higher than 140/80 mmHg despite use of antihypertensive drug(s) regularly
* Patients with chronic renal failure who need dialysis
* Patients who had prerenal, renal or postrenal acute kidney failure during the last 6 months
* Patients who had acute pyelonephritis during the last 6 months
* Patients younger than 18 years old or older than 65 years old
* Patients who had kidney surgery during the last 3 months and who have abnormal kidney functions
* Patients with ureteral stone who are planned to undergo endoscopic stone treatment at the same time
* Patients with a history of corticosteroid use during enrollment into the study or previous 3 months
* Patients with uncontrolled thyroid disease
* Patients who have a disease with rapid cell turn-over (like leukemia, lymphoma, etc.)
* Patients whose operation terminated or converted to open surgery due to any reason
* Patients with missing data

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-10-08 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Stone-free rate | Within the first 30 days after surgery.
  Determination of any residual stone in the collecting system by using one of imaging modalities.

SECONDARY OUTCOMES:
Complication rate | Within the first 30 days after surgery.
  Determination of any complications related to the surgery.
Blood Cystatin C level (mg/L) | Within the first 12 hours after surgery.
  Determination of any impairment in renal function after the surgery/procedure by measuring blood Cystatin C level.
Urine Cystatin C level (mg/L) | Within the first 12 hours after surgery.
  Determination of any impairment in renal function after the surgery/procedure by measuring urine Cystatin C level.

CONTACTS AND LOCATIONS:
Overall Officials: Ozcan Kilic, M.D., Principal Investigator — Selcuk University, School of Medicine, Department of Urology
Locations (1):
- Selcuk University, School of Medicine, Department of Urology, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de la Rosette J, Assimos D, Desai M, Gutierrez J, Lingeman J, Scarpa R, Tefekli A; CROES PCNL Study Group. The Clinical Research Office of the Endourological Society Percutaneous Nephrolithotomy Global Study: indications, complications, and outcomes in 5803 patients. J Endourol. 2011 Jan;25(1):11-7. doi: 10.1089/end.2010.0424. PMID 21247286
- [Background] Xu S, Shi H, Zhu J, Wang Y, Cao Y, Li K, Wang Y, Sun Z, Xia S. A prospective comparative study of haemodynamic, electrolyte, and metabolic changes during percutaneous nephrolithotomy and minimally invasive percutaneous nephrolithotomy. World J Urol. 2014 Oct;32(5):1275-80. doi: 10.1007/s00345-013-1204-2. Epub 2013 Nov 1. PMID 24177788
- [Background] Wong KA, Sahai A, Patel A, Thomas K, Bultitude M, Glass J. Is percutaneous nephrolithotomy in solitary kidneys safe? Urology. 2013 Nov;82(5):1013-6. doi: 10.1016/j.urology.2013.06.034. Epub 2013 Aug 16. PMID 23958507
- [Background] Kamphuis GM, Baard J, Westendarp M, de la Rosette JJ. Lessons learned from the CROES percutaneous nephrolithotomy global study. World J Urol. 2015 Feb;33(2):223-33. doi: 10.1007/s00345-014-1367-5. Epub 2014 Aug 7. PMID 25100624
- [Background] De S, Autorino R, Kim FJ, Zargar H, Laydner H, Balsamo R, Torricelli FC, Di Palma C, Molina WR, Monga M, De Sio M. Percutaneous nephrolithotomy versus retrograde intrarenal surgery: a systematic review and meta-analysis. Eur Urol. 2015 Jan;67(1):125-137. doi: 10.1016/j.eururo.2014.07.003. Epub 2014 Jul 23. PMID 25064687
- [Background] Bader MJ, Gratzke C, Seitz M, Sharma R, Stief CG, Desai M. The "all-seeing needle": initial results of an optical puncture system confirming access in percutaneous nephrolithotomy. Eur Urol. 2011 Jun;59(6):1054-9. doi: 10.1016/j.eururo.2011.03.026. Epub 2011 Apr 1. PMID 21477921
- [Background] Desai MR, Sharma R, Mishra S, Sabnis RB, Stief C, Bader M. Single-step percutaneous nephrolithotomy (microperc): the initial clinical report. J Urol. 2011 Jul;186(1):140-5. doi: 10.1016/j.juro.2011.03.029. Epub 2011 May 14. PMID 21575966
- [Background] Hatipoglu NK, Tepeler A, Buldu I, Atis G, Bodakci MN, Sancaktutar AA, Silay MS, Daggulli M, Istanbulluoglu MO, Karatag T, Gurbuz C, Armagan A, Caskurlu T. Initial experience of micro-percutaneous nephrolithotomy in the treatment of renal calculi in 140 renal units. Urolithiasis. 2014 Apr;42(2):159-64. doi: 10.1007/s00240-013-0631-2. Epub 2013 Dec 13. PMID 24337646
- [Background] Karatag T, Tepeler A, Buldu I, Akcay M, Tosun M, Istanbulluoglu MO, Armagan A. Is micro-percutaneous nephrolithotomy surgery technically feasible and efficient under spinal anesthesia? Urolithiasis. 2015 Jun;43(3):249-54. doi: 10.1007/s00240-015-0752-x. Epub 2015 Jan 9. PMID 25572955
- [Background] Desai J, Solanki R. Ultra-mini percutaneous nephrolithotomy (UMP): one more armamentarium. BJU Int. 2013 Nov;112(7):1046-9. doi: 10.1111/bju.12193. Epub 2013 Jul 11. PMID 23841665
- [Background] Shlipak MG, Mattes MD, Peralta CA. Update on cystatin C: incorporation into clinical practice. Am J Kidney Dis. 2013 Sep;62(3):595-603. doi: 10.1053/j.ajkd.2013.03.027. Epub 2013 May 20. PMID 23701892
- [Background] Delanaye P, Cavalier E, Morel J, Mehdi M, Maillard N, Claisse G, Lambermont B, Dubois BE, Damas P, Krzesinski JM, Lautrette A, Mariat C. Detection of decreased glomerular filtration rate in intensive care units: serum cystatin C versus serum creatinine. BMC Nephrol. 2014 Jan 13;15:9. doi: 10.1186/1471-2369-15-9. PMID 24410757
- [Background] Krawczeski CD, Vandevoorde RG, Kathman T, Bennett MR, Woo JG, Wang Y, Griffiths RE, Devarajan P. Serum cystatin C is an early predictive biomarker of acute kidney injury after pediatric cardiopulmonary bypass. Clin J Am Soc Nephrol. 2010 Sep;5(9):1552-7. doi: 10.2215/CJN.02040310. Epub 2010 Jun 10. PMID 20538834